CLINICAL TRIAL: NCT03564210
Title: The Effect of Screen Time on Recovery From Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodore Macnow (Other)
Responsible Party: Sponsor-Investigator, Theodore Macnow, Assistant professor of pediatrics, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H00014355
Record Dates: First submitted 2018-05-23; First posted 2018-06-20 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Concussion, Brain
Keywords: screen time
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screen time permitted (Active Comparator): Concussion sufferers permitted screen time for first 48 hours of recovery
  Interventions: Behavioral: Screen time permitted
- Screen time abstain (Active Comparator): Concussion sufferers asked to abstain from screen time for first 48 hours of recovery
  Interventions: Behavioral: Screen Time Abstain

INTERVENTIONS:
Behavioral: Screen time permitted — Cohort will not be directed to abstain from screen time
  Arms: Screen time permitted
Behavioral: Screen Time Abstain — Cohort will be directed to abstain from screen time
  Arms: Screen time abstain

SUMMARY:
This study will prospectively examine the effect of screen time on recovery from concussion. Patients 12 to 25 years of age presenting to the ED with a concussion will be randomized to allow for screen time as tolerated or to abstain from screen time for the first 48 hours of recovery. The amount of screen time use and duration of concussive symptoms will be assessed through daily surveys and a daily post-concussive symptom score (PCSS).

ELIGIBILITY:
Inclusion Criteria:

* Individuals presenting to the emergency department with a traumatic head injury sustained in the last 24 hours and diagnosed concussion as defined by Acute Concussion Evaluation tool (ACE-ED)
* Between 12 and 25.99 years of age
* English-speaking
* Subject (and parent/guardian when applicable) is able and willing to provide informed consent and assent
* pregnant women,

Exclusion Criteria:

* individuals who have a Glasgow Coma Scale score of 13 or less;
* have brain abnormalities on imaging;
* have severe preexisting neurological conditions;
* a concussion diagnosed within the last 2 weeks;
* have significant developmental delay;
* are intoxicated;
* require neurosurgical intervention, intubation, or hospital admission
* individuals who do not meet the age criteria;
* non-English speaking;
* prisoners;
* unable or unwilling to provide informed consent;
* Are under the age of 18 and do not have a parent/guardian with them who is willing and able to consent.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Duration of concussive symptoms | From date of randomization until PCSS of less than 7 is achieved or up to 10 days, whichever comes first.
  The average number of days from initial concussion diagnosis until participant has a Post Concussive Symptom Scale Score (PCSS) of less than 7

SECONDARY OUTCOMES:
Number of specific symptoms (Day 1-3) | Day 1 to day 3
  The average total number of symptoms as reported on the Post Concussive Symptom Scale (PCSS) by participant.
Number of specific symptoms each day (Day 4-10) | Day 4 to day 10
  The average total number of symptoms as reported on the Post Concussive Symptom Scale (PCSS) by participant.
Severity of specific symptoms (Day 1-3) | Day 1 to day 3
  The average severity of symptoms as reported on the Post Concussive Symptom Scale (PCSS) by participant.
Severity of specific symptoms (Day 4-10) | Day 4 to day 10
  The average severity of symptoms as reported daily by participant on the Post Concussive Symptom Scale (PCSS) by participant.
Amount of screen time use | Randomization to 48 hours.
  Average minutes of screen time (video games, television, computer, smartphone) as self-reported by participant on questionnaire.
Days until return to school/work and sports | From date of randomization to return to school/work and sports, up to day 10.
  The average number of days until the participant is able to return to routine activities such as school/work and sports as self-reported on questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Macnow, MD, Principal Investigator — UMass Memorial Health
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macnow T, Curran T, Tolliday C, Martin K, McCarthy M, Ayturk D, Babu KM, Mannix R. Effect of Screen Time on Recovery From Concussion: A Randomized Clinical Trial. JAMA Pediatr. 2021 Nov 1;175(11):1124-1131. doi: 10.1001/jamapediatrics.2021.2782. PMID 34491285